CLINICAL TRIAL: NCT00223483
Title: Identification and Analysis of Immunomodulatory Molecules From Leukocytes in Patients With Hematologic Disorders and Healthy Volunteers
Brief Title: Identification and Analysis of Immunomodulatory Molecules in Patients With Hematologic Disorders and Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: HSC20040268H
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Hematologic Diseases; Healthy Volunteers
Keywords: Hematologic Diseases; Genomics; Cytokines; Chemokines; Receptors
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, white cells
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Isolation of genomic DNA — One time blood draw

SUMMARY:
This research study goal is to analyze the plasma and the cells that make up part of the immune system. We want to learn how the plasma and cells work. These may influence why one person will develop an infection and another will not, or why one person develops severe symptoms of a disease while others remain without symptoms.

DETAILED DESCRIPTION:
This research study goal is to analyze the plasma and the cells that make up part of the immune system. These cells, called white cells or leukocytes, are present in blood. We want to learn how these cells work to prevent infection and how they respond after an infection occurs. We also want to study certain molecules present on the plasma, on or in these cells, and the genetic material that allows these molecules to be made. These molecules may influence why one person will develop an infection and another will not, or why one person develops severe symptoms of a disease while others remain without symptoms. This study may increase our understanding of a variety of diseases including infections such as HIV, allergic diseases such as asthma, joint diseases such as rheumatoid arthritis, certain cancers, and the rejection process that sometimes occurs after transplantation of an organ.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to give blood
* Must be able to give informed consent
* Signed, written informed consent

Exclusion Criteria:

* Individuals with a history severe anemia, inadequate venous access, severe blood or coagulation disorders.
* Pregnant women are excluded because it is a unique immunotolerant state and will alter the profile of immunomodulatory molecules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic and community samples
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2005-03; Primary Completion 2020-12-11 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Repository collection of plasma and serum for future analysis. | 12 years

CONTACTS AND LOCATIONS:
Overall Officials: Cesar O Freytes, MD, Study Director — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Department of Veterans Affairs, South Texas Veterans Health Care System, Audie L. Murphy Memorial Veterans Hospital Division, San Antonio, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas